CLINICAL TRIAL: NCT00041314
Title: A Phase II Trial Of Carboplatin And Gemcitabine With Exisulind In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069467; E-E1501
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; sulindac sulfone; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: exisulind
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of carboplatin, gemcitabine, and exisulind in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 18-month survival rate in patients with advanced non-small cell lung cancer treated with carboplatin, gemcitabine, and exisulind.
* Determine the feasibility and toxicity of this regimen in these patients.
* Determine the response rate, progression-free survival, and overall median survival of patients treated with this regimen.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Chemotherapy repeats every 21 days for up to 6 courses. Patients also receive oral exisulind twice daily beginning on day 1 of course 1 and continuing until disease progression or unacceptable toxicity occurs.

Patients are followed every 3 months for 2 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Unresectable stage IIIB (e.g., pleural effusion) not suitable for combined modality therapy OR
  * Stage IV
* Prior brain metastases are allowed provided the following are true:

  * Patient completed radiotherapy and/or surgery at least 3 weeks prior to study
  * Objective evidence of resolution or significant improvement of brain lesions exists on follow-up CT scan or MRI
  * Patient is neurologically improved or stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* WBC at least 3,000/mm^3
* Hemoglobin at least 9 g/L
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 mg/dL
* SGOT no greater than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No prior uncontrolled cardiovascular disease
* No hospitalization for acute myocardial infarction, arrhythmia, or congestive heart failure within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No serious active infection
* No dementia or active psychoses
* No other prior malignancy except nonmetastatic nonmelanoma skin cancer, carcinoma in situ of the cervix, or cancer curatively treated with surgery or small-field radiotherapy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 1 month since prior investigational agents
* More than 7 days since prior aspirin, sulindac, cyclo-oxygenase-2 (COX-2) inhibitors, or nonsteroidal anti-inflammatory drugs (except ibuprofen or naproxen)
* No concurrent sulindac or COX-2 inhibitors

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10-04 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2007-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Masters, MD, Study Chair — Endeavor Health
Locations (79):
- United States (75):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Burgess Health Center, Onawa, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- NSW Breast Cancer Institute, Westmead, New South Wales, Australia
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Masters GA, Li S, Dowlati A, Madajewicz S, Langer C, Schiller J, Johnson D. A phase II trial of carboplatin and gemcitabine with exisulind (IND #65,056) in patients with advanced non-small cell lung cancer: an Eastern Cooperative Oncology Group study (E1501). J Thorac Oncol. 2006 Sep;1(7):673-8. PMID 17409935